CLINICAL TRIAL: NCT00405353
Title: Testosterone Treatment for Multiple Sclerosis: A Preliminary Trial
Brief Title: Testosterone Treatment for Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Rhonda Voskuhl, Professor, Department of Neurology; Director Multiple Sclerosis Program, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG 3239
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; testosterone
MeSH Terms: conditions — Multiple Sclerosis | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- crossover treatment with Androgel (Experimental): 6 months pretreatment, 12 months treatment intervention with Androgel 10 grams of gel containing 100mg of testosterone
  Interventions: Drug: Androgel 10 grams of gel containing 100 mg of testosterone

INTERVENTIONS:
Drug: Androgel 10 grams of gel containing 100 mg of testosterone — testosterone gel
  Other Names: testosterone

SUMMARY:
Since men are less likely to develop multiple sclerosis, the hypothesis was that testosterone might be protective in MS. Men with MS for followed untreated for 6 months, followed by a 12 month treatment period with Androgel.

DETAILED DESCRIPTION:
Background: Men are less susceptible to many autoimmune diseases including multiple sclerosis (MS). Possible causes for this include sex hormones and/or sex chromosome effects. Testosterone treatment ameliorates experimental allergic encephalomyelitis (EAE), an animal model of MS, but the effect of testosterone supplementation on men with MS is not known.

Design, Setting and Participants: Ten men with relapsing remitting MS were studied using a crossover design whereby each patient served as his own control. There was a six-month pretreatment period followed by a twelve month period of daily treatment with 100mg of testosterone gel.

Main Outcome Measures: Brain atrophy and Cognitive testing

ELIGIBILITY:
Inclusion Criteria:

1. Men, age 18-65, with a diagnosis of clinically definite relapsing remitting multiple sclerosis.
2. Relapsing remitting patients who have declined or not tolerated treatment with beta interferon (Betaseron, Avonex) or glatiramer acetate, copolymer-1 (Copaxone).
3. At least one relapse in the two years prior to entry. Relapse will be defined historically as definite worsening of a previous symptom (over 0-3 days) or development of a new symptom (over 0-3 days).
4. Not in an intercurrent relapse.
5. Expanded Disability Status Score (EDSS) = 0.0 to 5.0.
6. The patients must have a significant T2 burden of disease on screening cerebral MRI as defined by T2 lesion loads greater than 7.5cm3.
7. Must live within 100 miles of UCLA.
8. Must be willing and able to receive an initial screening cerebral MRI, a baseline MRI and monthly cerebral MRIs (with and without gadolinium) for a total period of 12 months (6 months prior to treatment and 6 months during treatment).

Exclusion Criteria:

1. Males unable to fulfill the above criteria and all female patients.
2. Males who have been on sex hormone treatment including androgens, estrogens, or anti-estrogens for hypogonadism or other medical condition during the 12 months prior to study.
3. Males who have taken DHEA during the 3 months prior to study.
4. Patients who have thrombosis, serious cardiac, pulmonary, renal, gastrointestinal, hepatic, immunologic, infectious, neoplastic (with particular focus on patients with known or suspected estrogen or testosterone-dependent tumors), or urologic disease (with a particular focus on patients with a history of prostatic hypertrophy/nodules).
5. Patients with an abnormal prostate as evidenced by prostatic masses or induration on rectal examination or prostate ultrasonography or elevated levels of prostatic specific antigen (PSA 4 ng/ml or higher).
6. Patients with testicular mass on exam.
7. Patients with hematocrit greater than 50%
8. Patients with major psychiatric illness (e.g. manic depressive states, schizophrenia)
9. Patients with active alcoholism.
10. Patients with a history of drug abuse within the past five years.
11. Patients who are greater than 130% or less than 80% of their ideal body weight based on Metropolitan Life Tables.
12. Patients with generalized skin disease that may effect absorption of testosterone (e.g. psoriasis) or a known skin intolerance to alcohol.
13. Patients with prolactin > 40 mcg/L.
14. Patients with a cholesterol level greater than 300 mg/dl.
15. Patients with other conditions that would interfere with assessing neurologic functions such as deforming arthritis or a major amputation.
16. Patients who have received treatment with beta interferon (Betaseron or Avonex), glatiramer acetate copolymer-1 (Copaxone), ACTH, corticosteroids, intravenous immunoglobulins (IVIG), or plasma exchange in the three months preceding enrollment
17. Patients who have received treatment with azathioprine, cyclophosphamide, methotrexate, mitoxantrone, cyclosporin A or experimental therapies in the six months preceding enrollment.
18. Patients who have been treated with total lymphoid irradiation, monoclonal antibody, T cell vaccination, cladribine or bone marrow transplantation.
19. Patients who have positive titers to HIV1,2; HTLV1; or VDRL.
20. Patients who have clinical evidence of Lyme disease.
21. Patients who are mentally or emotionally incompetent in the opinion of the examining neurologist or unable to give informed consent, or to understand and comply with the study protocol.
22. Patients with certain artificial heart valves, pacemakers, or other metallic/electronic material in their bodies.
23. Patients with known hypersensitivity to gadolinium-DPTA.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Voskuhl, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziehn MO, Avedisian AA, Dervin SM, Umeda EA, O'Dell TJ, Voskuhl RR. Therapeutic testosterone administration preserves excitatory synaptic transmission in the hippocampus during autoimmune demyelinating disease. J Neurosci. 2012 Sep 5;32(36):12312-24. doi: 10.1523/JNEUROSCI.2796-12.2012. PMID 22956822
- [Result] Sicotte NL, Giesser BS, Tandon V, Klutch R, Steiner B, Drain AE, Shattuck DW, Hull L, Wang HJ, Elashoff RM, Swerdloff RS, Voskuhl RR. Testosterone treatment in multiple sclerosis: a pilot study. Arch Neurol. 2007 May;64(5):683-8. doi: 10.1001/archneur.64.5.683. PMID 17502467
- [Result] Gold SM, Chalifoux S, Giesser BS, Voskuhl RR. Immune modulation and increased neurotrophic factor production in multiple sclerosis patients treated with testosterone. J Neuroinflammation. 2008 Jul 31;5:32. doi: 10.1186/1742-2094-5-32. PMID 18671877
- [Result] Kurth F, Luders E, Sicotte NL, Gaser C, Giesser BS, Swerdloff RS, Montag MJ, Voskuhl RR, Mackenzie-Graham A. Neuroprotective effects of testosterone treatment in men with multiple sclerosis. Neuroimage Clin. 2014 Mar 6;4:454-60. doi: 10.1016/j.nicl.2014.03.001. eCollection 2014. PMID 24634831

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone Arm/ Group: All subjects underwent a 6-month observation period, followed by 12 months of open label testosterone treatment, using 10g of gel containing 100mg of testosterone (Androgel) applied topically.
Period: Overall Study
Arm/Group | Testosterone Arm/ Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Testosterone Arm/ Group: All subjects underwent a 6-month observation period, followed by 12 months of open label testosterone treatment, using 10g of gel containing 100mg of testosterone (Androgel) applied topically. Brain MRIs were obtained every month from baseline (month 0) until the end of the trial (month 18). All 10 subjects completed all nineteen monthly scans.
Arm/Group | Testosterone Arm/ Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex/Gender, Customized [Number; unit: patients]
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Whole Brain Atrophy Rate
Description: as assessed by Voxel-Based Morphometry
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: percent change in brain volume
Arm/Group | Testosterone Arm/ Group
Number analyzed (Participants) | 10
percent change in brain volume | .82 [.78 to .84]
Statistical Analysis 1: Comparison: Testosterone Arm/ Group; Percent change in brain volume against time scatter plot with a Loess regression curve was produced and a first-degree spline model was developed. This model fitted line pieces for pre-treatment and early treatment periods (month -6 to month 3) and treatment response period (months 3-12), and these pieces were joined together to achieve continuity. Slopes of these lines were estimated and compared. A random intercept was set in the model to allow the difference among subjects; Test type: Other; p < 0.05, Mixed Models Analysis; Linear regressions were used to determine slopes of brain volume changes. Statistical software package SAS was used to perform the analysis

ADVERSE EVENTS:
Time Frame: 18 months
Description: All subjects underwent a 6-month observation period, followed by 12 months of open label testosterone treatment, using 10g of gel containing 100mg of testosterone (Androgel) applied topically.
Arm/Group | Testosterone Arm/ Group
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No